CLINICAL TRIAL: NCT03233711
Title: A Randomized Phase III Study of Nivolumab After Combined Modality Therapy (CMT) in High Risk Anal Cancer
Brief Title: Nivolumab After Combined Modality Therapy in Treating Patients With High Risk Stage II-IIIB Anal Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01347; NCI-2017-01347 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA2165 (Other: ECOG-ACRIN Cancer Research Group); EA2165 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2017-07-28; First posted 2017-07-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Anal Basaloid Carcinoma; Anal Canal Cloacogenic Carcinoma; Anal Margin Squamous Cell Carcinoma; Stage IIB Anal Cancer AJCC v8; Stage III Anal Cancer AJCC v8
MeSH Terms: conditions — Anal Canal Carcinoma; Anus Neoplasms | interventions — Biopsy; Specimen Handling; Colonoscopy; Magnetic Resonance Spectroscopy; Nivolumab; Watchful Waiting; Observation; Proctoscopy; Sigmoidoscopy; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (nivolumab) (Experimental): Patients receive nivolumab while on study. Patients undergo sigmoidoscopy, colonoscopy or anoscopy, proctoscopy or digital rectal exam, x-ray, CT scan, MRI, biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Colonoscopy; Procedure: Computed Tomography; Procedure: Digital Rectal Examination; Procedure: High Resolution Anoscopy; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Proctoscopy; Procedure: Sigmoidoscopy; Procedure: X-Ray Imaging
- Arm B (clinical observation) (Other): Patients undergo observation while on study. Patients undergo sigmoidoscopy, colonoscopy or anoscopy, proctoscopy or digital rectal exam, x-ray, CT scan, MRI, biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Colonoscopy; Procedure: Computed Tomography; Procedure: Digital Rectal Examination; Procedure: High Resolution Anoscopy; Procedure: Magnetic Resonance Imaging; Other: Patient Observation; Procedure: Proctoscopy; Procedure: Sigmoidoscopy; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Arm A (nivolumab)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Colonoscopy — Undergo colonoscopy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Digital Rectal Examination — Undergo digital rectal examination
  Other Names: DRE
Procedure: High Resolution Anoscopy — Undergo anoscopy
  Other Names: HRA
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm A (nivolumab)
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Arm B (clinical observation)
Procedure: Proctoscopy — Undergo proctoscopy
Procedure: Sigmoidoscopy — Undergo sigmoidoscopy
  Other Names: Proctosigmoidoscopy
Procedure: X-Ray Imaging — Undergo chest x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase III trial investigates how well nivolumab after combined modality therapy works in treating patients with high risk stage II-IIIB anal cancer. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether therapy with nivolumab following combined modality therapy (CMT) improves disease-free survival (DFS) compared with observation in patients with high risk anal carcinoma.

SECONDARY OBJECTIVES:

I. To compare nivolumab following combined modality therapy (CMT) with observation in patients with high risk anal carcinoma with regard to:

Ia. Objective response rate (complete [CR] and partial [PR]), stable disease and progression.

Ib. Severe toxicity interval. Ic. Colostomy-free survival. Id. Overall survival. Ie. Toxicity.

OUTLINE: Patients who received standard CMT are randomized to 1 of 2 arms.

ARM A: Patients receive nivolumab intravenously (IV) while on study.

ARM B: Patients undergo observation while on study

Patients undergo sigmoidoscopy, colonoscopy or anoscopy, proctoscopy or digital rectal exam, x-ray, computed tomography (CT) scan, magnetic resonance imaging (MRI), biopsy and blood sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Age >= 18 years
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Patients must have histologically proven stage IIB (T3N0M0 only), IIIA (T2N1M0), IIIB (T4N0M0), or IIIC (T3N1M0, T4N1M0) invasive squamous cell carcinoma of the anus or anorectum, according to the American Joint Committee on Cancer (AJCC) 8th edition; this may include tumors of non-keratinizing histology such as basaloid, transitional cell, or cloacogenic histology; individuals with squamous cell carcinoma of the anal margin are eligible if there is evidence of extension of the primary tumor into the anal canal
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Patients must have hemoglobin levels of > 9 g/dL (within 2 weeks prior to registration)
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Patient must have a platelet count of > 100,000/mm^3 (within 2 weeks prior to registration)
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Patient's absolute neutrophil count (ANC) level must be > 1500/mm^3 (within 2 weeks prior to registration)
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Serum creatinine must be =< 1.5 X upper limit of normal (ULN) (within 2 weeks prior to registration)
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Total bilirubin must be < 2 X ULN (within 2 weeks prior to registration)
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X institutional upper limit of normal (within 2 weeks prior to registration)
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Albumin >= 3.0 g/dL (within 2 weeks prior to registration)
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Patients known to be human immunodeficiency virus (HIV)+ are permitted; patients with CD4 > 200 and serum HIV viral load of < 200 copies/mm^3 are eligible, and in addition:

  * Participants must be purified protein derivative (PPD) negative; alternatively, the QuantiFERON-tuberculosis (TB) Gold In-Tube (QFT-GIT) assay (Cellestis Limited, Carnegie, Australia) can be used; an individual is considered positive for M. tuberculosis infection if the IFN-gamma response to TB antigens is above the test cut-off (after subtracting the background IFN-gamma response in the negative control); the result must be obtained within 20 weeks prior to enrollment; PPD positive (or Quantiferon assay positive) participants are permitted if prophylaxis has been completed prior to enrollment
  * No history of acquired immune deficiency syndrome (AIDS)-related complications within past year other than a history of low CD4+ T-cell count > 200/mm^3 prior to initiation of combination antiretroviral therapy; on study CD4+ T-cell count may not be informative due to chemoradiotherapy and should not be used as an exclusion criterion if low
  * Patient must be healthy on the basis of HIV disease with high likelihood of near normal life span were it not for the anal cancer
  * Participants MUST receive appropriate care and treatment for HIV infection, including antiretroviral medications when clinically indicated, and should be under the care of a physician experienced in HIV management; participants will be eligible regardless of antiretroviral medication (including no antiretroviral medication) provided there is no intention to initiate therapy or the regimen has been stable for at least 4 weeks with no intention to change the regimen within 12 weeks following enrollment
  * Patient must have =< grade 2 diarrhea (participants with grade 1 diarrhea are eligible provided stool for ova/parasites and stool cryptosporidium studies are negative;
  * NOTE: HIV testing is not required for eligibility
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: For patients registering prior to start of chemoradiotherapy, baseline scans must have been completed within 4 weeks prior to registration
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Women of child bearing potential and sexually active males must use accepted and effective method(s) of contraception and/or abstain from sexual intercourse while on protocol treatment and for at least 5 months after the last dose of nivolumab (for female patients) and for at least 7 months after the last dose of nivolumab (for male patients)
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Any surgery must have been completed >= 4 weeks prior to starting study treatment
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: No uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: No prior treatment with an immune checkpoint inhibitor (anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4 monoclonal antibody)
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: No patients with immunodeficiency or receiving systemic steroid therapy equivalent to > 10 mg prednisone per day or any other form of immunosuppressive therapy within 7 days prior to Step 1 registration; topical corticosteroid or occasional inhaled corticosteroids are allowed
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: No live vaccines within 30 days prior to registration; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccine; seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines and are not allowed

  * NOTE: no live vaccines may be administered while participating in the trial
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Previously irradiated patients (Arm S) must have received radiation per National Comprehensive Cancer Network guidelines; radiation therapy delivered on protocol (Arm T) will be reviewed
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patients will be registered within 63 days following completion of standard chemoradiation for anal cancer; standard chemoradiation therapy is as defined
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patients must have histologically proven stage IIB (T3N0M0 only), IIIA (T2N1M0), IIIB (T4N0M0), or IIIC (T3N1M0, T4N1M0) invasive squamous cell carcinoma of the anus or anorectum, according to the AJCC 8th edition; this may include tumors of non-keratinizing histology such as basaloid, transitional cell, or cloacogenic histology; individuals with squamous cell carcinoma of the anal margin are eligible if there is evidence of extension of the primary tumor into the anal canal
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patients must have received at least 54 gray (Gy) of radiation to the PTVp (primary) and 45 Gy to PTVn (elective nodal region) for the treatment of the anal cancer
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patients must have ECOG performance status of 0-2
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patients must have hemoglobin levels of > 10 g/dL (within 2 weeks prior to registration)
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patient must have a platelet count of > 100,000/mm^3 (within 2 weeks prior to registration)
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patient's ANC level must be > 1500/mm^3 (within 2 weeks prior to registration)
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Serum creatinine must be =< 1.5 X ULN (within 2 weeks prior to registration)
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Total bilirubin must be < 2 X ULN (within 2 weeks prior to registration)
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: AST (SGOT)/ALT (SGPT) =< 2.5 X institutional upper limit of normal (within 2 weeks prior to registration)
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Albumin >= 3.0 g/dL (within 2 weeks prior to registration)
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patients known to be human immunodeficiency virus (HIV)+ patients with CD4 > 200 and serum HIV viral load of < 200 copies/mm^3 are eligible; in addition:

  * Participants must be PPD negative; alternatively, the QuantiFERON-TB Gold In-Tube (QFT-GIT) assay (Cellestis Limited, Carnegie, Australia) can be used; an individual is considered positive for M. tuberculosis infection if the IFN-gamma response to TB antigens is above the test cut-off (after subtracting the background IFN-gamma response in the negative control); the result must be obtained within 20 weeks prior to enrollment; PPD positive (or Quantiferon assay positive) participants are permitted if prophylaxis has been completed prior to enrollment; NOTE: If patient completed chemoradiation on Step 1, PPD testing does not need to be performed again
  * No history of AIDS-related complications within past year other than a history of low CD4+ T-cell count > 200/mm^3 prior to initiation of combination antiretroviral therapy; on study CD4+ T-cell count may not be informative due to chemoradiotherapy should not be used as an exclusion criterion if low
  * Patient must be healthy on the basis of HIV disease with high likelihood of near normal life span were it not for the anal cancer
  * Participants MUST receive appropriate care and treatment for HIV infection, including antiretroviral medications when clinically indicated, and should be under the care of a physician experienced in HIV management; participants will be eligible regardless of antiretroviral medication (including no antiretroviral medication) provided there is no intention to initiate therapy or the regimen has been stable for at least 4 weeks with no intention to change the regimen within 12 weeks following enrollment
  * Patient must have =< grade 2 diarrhea (participants with grade 1 diarrhea are eligible provided stool for ova/parasites and stool cryptosporidium studies are negative)
  * NOTE: HIV testing is not required for eligibility
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Scans done within 4 weeks of randomization to Step 2
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patient must have recovered from all toxicities associated with chemoradiotherapy for anal cancer, to grade =< 1 with the exception of alopecia
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Women of child bearing potential and sexually active males must use accepted and effective method(s) of contraception and/or abstain from sexual intercourse while on protocol treatment and for at least 5 months after the last dose of nivolumab (for female patients) and for at least 7 months after the last dose of nivolumab (for male patients)
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: No uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: No prior treatment with an immune checkpoint inhibitor (anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4 monoclonal antibody)
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: No patients with immunodeficiency or receiving systemic steroid therapy equivalent to > 10 mg prednisone per day or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication; topical corticosteroid or occasional inhaled corticosteroids are allowed
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: No live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccine; seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines and are not allowed

Exclusion Criteria:

* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: For patients registering to Arm T, patients must not have received prior chemoradiotherapy for anal cancer
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Patients with an allogenic bone marrow/stem, cell or solid organ transplant are excluded
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Women MUST NOT be pregnant or breast-feeding due to the potential teratogenic harm or abortifacient effects to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used; all patients must also not expect to conceive or father children from study registration and throughout their time on study treatment; for female patients this must continue until at least 5 months after the last dose of nivolumab and for male patients until at least 7 months after the last dose of nivolumab; all females of child bearing potential must have a serum or urine pregnancy test to rule out pregnancy within 2 weeks prior to registration; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Patients will be excluded if they have a T1 or M1, and T2N0 cancer
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Patients must not have had prior potentially curative surgery (abdominal, peritoneal resection) for carcinoma of the anus
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Participants may not be receiving any other standard anti-cancer therapy or experimental agent concurrently with the study drugs
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Individuals with a history of a different malignancy are ineligible except if they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence; individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Patient must not have active autoimmune disease in the past 2 years

  * NOTE: This does not include patients with autoimmune disease controlled by medication, such as hypothyroidism; this eligibility includes only patients with endocrine disease controlled by hormone replacement, e.g. hypothyroid, adrenal insufficiency, or diabetes mellitus (DM)
* REGISTRATION TO STEP 1 ELIGIBILITY CRITERIA: Patients must not have known interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patients with an allogenic bone marrow/stem, cell or solid organ transplant are excluded
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Women MUST NOT be pregnant or breast-feeding due to the potential teratogenic harm or abortifacient effects to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used; all patients must also not expect to conceive or father children from study registration and throughout their time on study treatment; for female patients this must continue until at least 5 months after the last dose of nivolumab and for male patients until at least 7 months after the last dose of nivolumab; all females of child bearing potential must have a serum or urine pregnancy test to rule out pregnancy within 2 weeks prior to registration; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patients must not have had prior potentially curative surgery (abdominal, peritoneal resection) for carcinoma of the anus
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Participants may not be receiving any other standard anti-cancer therapy or experimental agent concurrently with the study drugs
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Individuals with a history of a different malignancy are ineligible except if they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence; individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patient must not have active autoimmune disease that has required systemic treatment in past 2 years
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patients must not have known interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* REGISTRATION TO STEP 2 ELIGIBILITY CRITERIA: Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2018-07-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | Up to 5 years
  Will be defined as the occurrence of progression of local disease, distant metastases, second primary or death from the date of randomization.

SECONDARY OUTCOMES:
Objective response rate | Up to 5 years
  Will be defined by complete and partial response.
Severe toxicity interval | The time between randomization and the occurrence of late severe side effects (up to 5 years)
  The following late side effects are considered as severe: any anal/rectal damage (ulcer, fistula, or perforation), rectal stenosis that required colostomy, skin ulceration, and severe fibrosis. This parameter estimates the probability of being free of late side effects for patients under loco-regional control.
Colostomy-free survival | Up to 5 years
Overall survival | Up to 5 years
Incidence of toxicities | Up to 5 years
  Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Rajdev, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (899):
- United States (890):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Enloe Medical Center, Chico, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Mills Health Center, San Mateo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - AdventHealth Celebration, Celebration, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Medical Group Urology at Orlando, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Franciscan Saint Elizabeth Health - Lafayette East, Lafayette, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Baptist Health Floyd, New Albany, Indiana
  - Union Hospital, Terre Haute, Indiana
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - McLaren Cancer Institute-Bloomfield, Bloomfield, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Hematology Oncology Consultants PC-Royal Oak, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Covenant HealthCare Mackinaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Wake Forest University at Elkin, Elkin, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Wake Forest University at Lexington, Lexington, North Carolina
  - Atrium Health Lincoln/LCI-Lincolnton, Lincolnton, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Wake Forest University at Mount Airy, Mount Airy, North Carolina
  - Rex Hematology Oncology Associates-Blue Ridge, Raleigh, North Carolina
  - UNC Health Cancer Care Raleigh, Raleigh, North Carolina
  - UNC Health Cancer Care Wakefield, Raleigh, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Sovah Health Martinsville, Martinsville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (9):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Algoma District Cancer Program Sault Area Hospital, Sault Ste. Marie, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan